CLINICAL TRIAL: NCT06005870
Title: Zanubrutinib Combined With Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone in the Treatment of Newly Diagnosed Diffuse Large B-cell Lymphoma With p53 Protein Expression
Brief Title: Zanubrutinib Combined With R-CHOP in the Treatment of Newly Diagnosed DLBCL With p53 Protein Expression
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Liling Zhang, Professor, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHCT22242
Record Dates: First submitted 2023-07-24; First posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: DLBCL; Diffuse Large b-cell lymphoma; p53; zanubrutinib
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — zanubrutinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Z-RCHOP (Experimental): Patients with newly diagnosed DLBCL with p53 expression were treated with a combination of Zanubrutinib and RCHOP.
  Interventions: Drug: Zanubrutinib plus RCHOP

INTERVENTIONS:
Drug: Zanubrutinib plus RCHOP — Rituximab 375mg/m2 D1; cyclophosphamide 750mg/m2 D2; adriamycin 50 mg/m2 D2 vincristine 1.4mg/m(Max 2mg) D2; prednisone 100mg/d D2-6; Zanubrutinib 160 mg, the bid D1-21

SUMMARY:
This study aim to evaluate the efficacy and safety of zanubrutinib combined with R-CHOP in the treatment of DLBCL patients with p53 protein expression.

DETAILED DESCRIPTION:
This is a prospective, single arm, single center study,it plans to recruit 41 newly diagnosed DLBCL patients with p53 protein expression(≥50%).According to Simon's two-stage optimal design criteria, 19 eligible patients were recruited in the first phase, and at least 12 patients were required to achieve complete response to enter the second phase. In phase 2, additional 22 patients were recruited. These patients will receive zanubrutinib plus RCHOP for 6 cycles. After 4 treatment cycles, an interim response assessment will be performed to evaluate disease progression for each participant. Participants with progressive or stable disease will be discontinued from treatment，Participants with complete/partial response will continue ZRCHOP until 6 cycles are completed.After completion of study drug, participants will undergo assessment of tumor response based on the Revised Response Criteria for Malignant Lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, ≤ 75 years, both sexes;
2. Diff use large B-cell lymphoma diagnosed by histopathology without previous systemic DLBCL treatment;
3. ECOG score: 0-2;
4. Predicted survival ≥3 months;
5. Patients with positive p53 expression detected by immunohistochemistry (≥50% );
6. The patients had certain conditions of organ function reserve, and the laboratory tests within 1 week before enrollment met the following conditions:

Blood routine: neutrophil count (NEUT) ≥1.5×10^9/L, platelet count (PLT)

≥75×10^9/L, hemoglobin (HGB) ≥80 g/L; G-CSF was not used in the past 7 days (the researchers judged that the lymphoma-induced cytopenia could be included).

Liver function: Total bilirubin (TBIL) ≤1.5× upper limit of the normal range (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN; If liver metastases were present, TBIL≤3×ULN, ALT and AST≤5×ULN; Renal function: serum creatinine (Cr) ≤2.0×ULN or creatinine clearance (CCr) ≥60ml/min;

Cardiac function: LVEF≥50%, ECG did not indicate any acute myocardial infarction, arrhythmia, or atrioventricular conduction block above grade I;

Thyroid function: thyroid stimulating hormone (TSH) was within the normal range. If TSH is abnormal, free triiodothyronine (FT3) and free thyroxine (FT4) should be within the normal range or abnormal without clinical significance.

1. According to the Lugano2014 assessment criteria, patients must have measurable lesions, defined as the longest diameter of at least one nodule > 1.5cm, or the longest diameter of at least one nodule > 1cm, and at least two vertical diameters that can be accurately measured.
2. Patients volunteered to participate in the trial, understood the study procedure, and were able to sign in-person informed consent.

Exclusion Criteria:

1. Patients with definite lymphoma central nervous system (CNS) infiltration, including brain parenchyma, meningeal invasion, or spinal cord compression;
2. severe or uncontrolled infection;
3. with active autoimmune disease;
4. Other serious medical conditions, such as uncontrolled diabetes, gastric ulcers, other serious cardiopulmonary diseases, etc. (the decision was left to the investigator);
5. patients who received the live attenuated vaccine within 4 weeks before the first dose or planned to receive the live attenuated vaccine during the study;
6. The subject has previous or co -e xis ting other malignant tumors; Patients with basal cell carcinoma of the skin and uterine and neck carcinoma in situ who had been cured for more than 3 years, and patients with other malignant tumors who had been cured for more than 5 years were considered for inclusion.
7. HIV-positive patients with active hepatitis B ( HBV-DNA > 100 copies/m L), positive HCV antibody, or abnormal HCV-RNA
8. Women who were pregnant or lactating, women who planned to become pregnant between the study period and 6 months after the last dose, or men whose partners planned to become pregnant, who were unwilling to use a medically approve defective contraceptive method (e.g., intrauterine device or condom ) during the trial;
9. were allergic to any of the drugs in the study protocol;
10. ineligible for inclusion as judged by the investigator ;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2022-11-26 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Complete response rate (CRR) | At the end of cycle 6 (each cycle is 21 days )
  To evaluate the efficacy of anti-lymphoma

SECONDARY OUTCOMES:
Overall response rate (ORR) | At the end of cycle 6 (each cycle is 21 days )
  To evaluate the efficacy of anti-lymphoma
Progression-free survival (PFS) | From date of initiation therapy until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  To evaluate the efficacy of anti-lymphoma
Overall survival (OS) | From date of initiation therapy until the date of death from any cause, assessed up to 60 months
  To evaluate the efficacy of anti-lymphoma
Rate of AE and SAE | from the initiation of the first dose to 28 days after the last dose
  To identify the incidence of AE and SAE in clinical trial

CONTACTS AND LOCATIONS:
Overall Officials: Liling Zhang, M.D, Study Chair — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China